CLINICAL TRIAL: NCT06935539
Title: A Prospective, Single-center, Open-label, Pilot Randomized Controlled Study Evaluating the Clinical Effectiveness of Lateral Branch Cryoneurolysis Versus Radiofrequency Ablation for the Treatment of Chronic Sacroiliac Joint Pain
Brief Title: Cryoneurolysis vs Radiofrequency Ablation for Chronic Sacroiliac Joint Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Pain Management Services, PLLC (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRS-131
Record Dates: First submitted 2025-04-10; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Chronic Sacroiliac Joint Pain
Keywords: low back pain; chronic low back pain; sacroiliac joint pain; chronic sacroiliac joint pain; cryoneurolysis; radiofrequency ablation
MeSH Terms: conditions — Low Back Pain | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Randomization to treatment groups according to the randomization assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cryoneurolysis (Active Comparator): Subjects will receive iovera° cryoneurolysis to the nerves of the sacroiliac joint
  Interventions: Device: Cryoneurolysis
- Radiofrequency ablation (Active Comparator): Subjects will receive RFA to nerves of the sacroiliac joint
  Interventions: Device: Radiofrequency ablation

INTERVENTIONS:
Device: Cryoneurolysis — The iovera° system consists of a reusable, portable Handpiece, along with single-patient use sterile Smart Tips (i.e., cryoprobes) and disposable nitrous oxide (N2O) cartridges. The iovera° system produces the desired effect through initiation of a cooling cycle. Each cooling cycle is initiated by fully inserting the Smart Tip into the selected procedure site and activating the cryogen flow. The Smart Tip needles are made of stainless steel and have a closed tip, fully enclosing the cryogen. The "STT21180STIM" Smart Tip will be used in this study.
  Other Names: iovera
  Arms: Cryoneurolysis
Device: Radiofrequency ablation — Radiofrequency ablation is a minimally invasive procedure that uses heat at the lumbosacral spine to destroy the target spinal nerves.
  Arms: Radiofrequency ablation

SUMMARY:
This is a single-center, randomized, open-label, pilot study in adult subjects with chronic sacroiliac joint (SIJ) pain. Thirty (30) subjects are planned for initial enrollment and will be randomized 1:1 to receive ioveraº cryoneurolysis or radiofrequency ablation.

DETAILED DESCRIPTION:
This is a single-center, randomized, pilot study in adult subjects with chronic SIJ pain. Thirty (30) subjects are planned for initial enrollment and will be randomized 1:1 to receive ioveraº cryoneurolysis or radiofrequency ablation (RFA).

This study is designed to evaluate the clinical effectiveness of iovera° cryoneurolysis in adult subjects with chronic SIJ pain. Furthermore, the study will assess the feasibility of the outcome measurements employed, construct a foundation for sample size calculation, and the acceptability/practicality of conducting an efficacy randomized controlled trial (RCT).

Randomization to treatment groups according to the randomization assignment will be performed on the day of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects at least 18 years of age at Screening
2. Primary complaint of buttock or axial low-back below L5 suggestive of unilateral or bilateral SIJ-mediated back pain
3. Positive SIJ provocative testing (at least two tests must be positive)

   1. Thigh thrust test
   2. Distraction test
   3. Gaenslen's test
   4. Compression test
   5. Sacral thrust test
4. Low back or buttock pain is chronic (i.e., ≥ 3 months' duration)
5. Low back or buttock pain is moderate to severe (score of ≥ 4 to ≤ 9) on the 0 to 10 NRS at Screening
6. Low back or buttock pain causes functional impairment (≥ 30% on ODI) at Screening
7. Successful trial of one diagnostic sacroiliac joint block with local anesthetic and steroids that results in at least 50% relief of primary (index) pain for the duration of the local anesthetic used
8. Failure of at least three months of conservative non-operative therapy (e.g., physical therapy, chiropractic care, sleep hygiene, weight loss, spinal injections, NSAIDs, physician-directed exercise program or other appropriate analgesics)
9. Able to provide informed consent, adhere to the study visit schedule, and complete all study assessment

Exclusion Criteria:

1. Active workers' compensation, personal injury, Social Security disability insurance (SSDI), or other litigation/compensation related to the spine
2. Serious spinal disorders (verified on magnetic resonance imaging (MRI)) that may impact outcomes, including any of the following:

   1. Suspected cauda equina syndrome (e.g., bowel/bladder dysfunction)
   2. Infection
   3. Tumor
   4. Traumatic fracture
   5. Systemic inflammatory spondyloarthropathy
   6. Lumbar radiculopathy/radiculitis (i.e., root irritation and deficit)
   7. Neurogenic claudication
3. Prior SIJ fusion surgery across the SI joint
4. Comorbidity that, in the judgment of the Investigator, may affect the subject's ability to participate in the study including lumbar radiculopathy and neuropathic pain disorder
5. Currently pregnant, nursing, or planning to become pregnant during the study
6. Known contraindication to study device, including any of the following:

   1. Cryoglobulinemia
   2. Paroxysmal cold hemoglobinuria
   3. Cold urticaria
   4. Raynaud's disease
   5. Open and/or infected wounds at or near the treatment site
   6. Coagulopathy
7. Previous participation in an iovera° study
8. Severe chronic pain disorder that in the opinion of the investigator may impact study outcomes
9. Presence of any of the following:

   1. Spinal neurostimulator
   2. Intrathecal analgesic drug pump
10. Current manifestation of poorly controlled mental illness or catastrophizing that in the opinion of the investigator may meaningfully impact treatment outcomes, including any of the following:

    a. Mood disorder (e.g., depression, bipolar) i. Patient Health Questionnaire (PHQ-9) ≥ 12 at Screening b. Psychotic disorder (e.g., schizophrenia) c. Catastrophizing i. Pain Catastrophizing Scale (PCS) score >30 at Screening
11. Subject received other spine interventions/therapies in the 30 days prior to block administration (e.g., spinal injections, minimally invasive therapies, surgical therapies) at the intended lumbar treatment levels
12. Subject received radiofrequency ablation ≤ 6 months before study enrollment at the intended treatment levels
13. History, suspicion, or clinical manifestation of:

    1. Alcohol abuse or dependence
    2. Illicit drug use
    3. Opioid abuse or dependence (≥40 mg MED PO/day in past 30 days) Given the COVID-19 pandemic, the subject must be medically fit/cleared for surgery by the investigator. If there is a concern about a subject's recent or potential exposure to COVID-19, or if the subject is not medically fit/cleared for surgery due to suspected COVID-19 illness/symptoms (or other serious illness), the subject must be excluded per Exclusion criterion #4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Safety and Clinical Effectiveness of Cryoneurolysis as Compared to Radiofrequency Ablation (RFA) | 0-12 months
  Safety will be assessed as the number of subjects with reported treatment-related adverse related to cryoneurolysis or RFA.

SECONDARY OUTCOMES:
Pain Intensity | 0-12 Months
  Subjects will evaluate their pain in the low back region using an 11-point Numeric Rating Scale (NRS), where 0=no pain and 10=worst possible pain.
  Subjects will evaluate how much pain they are currently experiencing and their average pain level over the past 24 hours.
Functional disability | 0-12 months
  Function disability will be measured by the Oswestry Disability Index. The score ranges from 0-50, with lower scores reflecting milder disability.
Concomitant medication use | 0-12 months
  Concomitant medication use will be collected per participant medication diary.
Success and failure rate of study interventions | Day 180
  Treatment success or failure will be determined at Day 180 (± 5 days) as described by Birkenmaier et al.:
  1. Full success of treatment is when pain is reduced to 50% or less of pre-treatment levels
  2. Partial success of treatment is when pain is reduced between 51-69% of pre-treatment levels
  3. Failure of treatment is when pain is reduced to 70% or greater of pre-treatment levels
Shor-form 12 (SF-12) | Screening, Day 90 (± 5 days), Day 180 (± 5 days), Day 270 (± 7 days), Day 360 (± 7 days)
  Health-related quality of life will be measured by the short-form (SF) 12. The SF-12 is a self administered 12-item questionnaire that assesses an individual's physical and mental health status across eight domains. Total scores range form 0-100 with scores above 50 indicating better-than-average health-related quality of life, and scores below 50 indicating below-average health.
Satisfaction With Pain Management | 12 months
  Subject satisfaction with pain management as measured on a scale ranging from 1) extremely dissatisfied 2) dissatisfied 3) neither satisfied nor dissatisfied 4) satisfied 5) extremely satisfied.
Patients' Global Impression of Change | 12 months
  The Patients' Global Impression of Change (PGIC) is an 11-point self-report scale assessing overall changes in activity limitations, symptoms, emotions, and quality of life, ranging from 0 to 10, where higher values indicate worse outcomes.

OTHER OUTCOMES:
Lost work days | 0-12 months
  Lost work days related to low back pain will be self-reported to evaluate the impact of cryoneurolysis on the number of lost workdays compared to radiofrequency ablation.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Ferrillo, DO, Principal Investigator — The Albany & Saratoga Centers For Pain Management

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Birkenmaier C, Veihelmann A, Trouillier H, Hausdorf J, Devens C, Wegener B, Jansson V, von Schulze Pellengahr C. Percutaneous cryodenervation of lumbar facet joints: a prospective clinical trial. Int Orthop. 2007 Aug;31(4):525-30. doi: 10.1007/s00264-006-0208-6. Epub 2006 Aug 23. PMID 16927087